CLINICAL TRIAL: NCT01186965
Title: Ehealth: Second Life Impacts Diabetes Education & Self-Management
Acronym: SLIDES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00022132; R21LM010727-02 (NIH)
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Second Life; virtual community; diabetes education; diabetes support group
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: eHealth program in the Virtual Environment (VE) platform Second Life — determine the feasibility and acceptability of an eHealth program that provides diabetes education and self-management support.
  Other Names: Second Life

SUMMARY:
The purpose of this study is to to develop and evaluate the feasibility, usability, and effect of participation in SLIDES (a virtual diabetes community in Second Life) for providing interactive diabetes education, support, and resources.

ELIGIBILITY:
Inclusion Criteria:

* current Duke Endocrinology patient
* are between 21 and 75 years old
* are able to speak and read English
* are computer literate (have used a computer for at least 6 months)
* understand how to use the Internet (have accessed the Internet on at least 6 occasions)
* have access to a computer with a non-dial-up Internet connection in a private location (home)
* are mentally capable of informed consent
* are reachable by telephone
* have no pre-existing medical condition(s) or severe diabetes related complications that would interfere with study participation (i.e., physical activity) or measures (e.g., renal failure, Stage III hypertension, severe orthopedic conditions or joint replacement scheduled within 6 months, paralysis, bleeding disorders, cancer, or receipt of pharmacologic doses of anti-coagulant medications [warfarin])
* are able to travel to Duke University Medical Center (DUMC) for follow-up appointments.

Exclusion Criteria:

-

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Perceived Usefulness | 3 and 6 months
Perceived Ease of Use | 3 and 6 months
Process data | January 2011 through May 2012

SECONDARY OUTCOMES:
Demographics | baseline
Metabolic Indicators | baseline, 3 months, 6 months
Diabetes knowledge | baseline, 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Constance M Johnson, PhD, Principal Investigator — Duke University School of Nursing
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States